CLINICAL TRIAL: NCT02443220
Title: Effects of Regional and Distant Combination of Acupoints Stimulated With Electroacupuncture on Patients Undergoing Off-pump Coronary Artery Bypass Grafting
Brief Title: Electroacupuncture in Reducing the Dose of Analgesic in Patients Undergoing Off-pump Coronary Artery Bypass Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, MD& PhD, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20140420-X-1; 81370011 (Other Grant/Funding Number: National nature and science foundation of China)
Record Dates: First submitted 2014-08-18; First posted 2015-05-13 (Estimated); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- distal-proximal group (Experimental): TEAS (transcutaneous electric acupoint stimulation) on "Danzhong" and "Hegu"
  Interventions: Device: TEAS (transcutaneous electric acupoint stimulation)
- regional group (Active Comparator): TEAS (transcutaneous electric acupoint stimulation) on "Danzhong" and "Juque"
  Interventions: Device: TEAS
- control group (Sham Comparator): no TEAS (transcutaneous electric acupoint stimulation) on "Danzhong" and "Hegu" .
  Interventions: Device: TEAS

INTERVENTIONS:
Device: TEAS (transcutaneous electric acupoint stimulation) — transcutaneous electric acupoint will commence at 30 min on "Danzhong" and "Hegu" before anesthesia in distal-proximal group
  Arms: distal-proximal group
Device: TEAS — transcutaneous electric acupoint will commence at 30 min on "Danzhong" and "Juque" before anesthesia in regional group
  Arms: regional group
Device: TEAS — The device will be connected to "Danzhong" and "Hegu" but no stimulation to the acupoints 30 min before anesthesia
  Arms: control group

SUMMARY:
A prospective, multiple-center, double-blinded, randomized, controlled clinical study to evaluate the antalgic effects between distal-proximal acupoints combination and regional acupoints combination stimulated with electroacupuncture on patients undergoing Off-Pump Coronary-Artery Bypass Grafting(OP-CABG).This clinical trial is to investigate whether electroacupuncture(EA) anesthesia can reduce analgesic in OP-CABG surgery in distal-proximal group.The origins of therapeutic acupuncture can be traced back at least 2,500 years in China. There has been an explosion of interest in Western medicine within the United States and Europe in application of acupuncture technique. Acupuncture enjoys worldwide acceptance for treating diseases such as migraine, chronic low back pain, and knee osteoarthritis. In 2002, WHO recommended 107 symptoms, syndromes, and diseases definitively shown to be effectively treated by acupuncture. Coronary heart disease (angina pectoris) is among these pathologies. A recent clinical trial demonstrated an acupuncture-assisted anesthesia strategy reduces postoperative morbidity and medical costs in open-heart surgery under cardiopulmonary bypass. Previous researches in animal models have demonstrated that electroacupuncture pretreatment protects the heart from ischemic injury. The investigators observed that electroacupuncture pretreatment (EAP, 30-minute electric stimulation through 4 electrodes attached to the bilateral forearm acupoints) before surgery significantly attenuated serum troponin levels during and shortly post-surgery in adult heart valve replacement patients and children undergoing cardiac surgery correcting congenital heart malformation.However, whether electroacupuncture anesthesia may reduce analgesic in OP-CABG surgery,especially in different combination of acupoints,has never been previously investigated.

DETAILED DESCRIPTION:
The anesthesia will be performed in a standard way. The propofol and sufentanil will be infused in target-controlled infusion mode. The dosage of analgesic will be assessed by the consumption of sufentanil. And the electroacupuncture anesthesia will be implemented by a device named "Hua Tuo" electronic acupuncture treatment instrument.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists I-III
* Scheduled for Off-Pump Coronary-Artery Bypass Grafting surgery
* First thoracotomy
* Signed written informed consent obtained

Exclusion Criteria:

* American Society of Anesthesiologists IV
* Undergoing surgery within 12 h of admission to hospital
* Life expectancy < 1 year at the time of enrollment
* Hemodynamic instability as defined by a systolic blood pressure <90 mmHg
* Preoperative Intra-aortic Balloon Pumping or Ventricular Assisted Device
* Severe hepatic or renal dysfunction
* Not the first thoracotomy
* Mediastinal fiber thickening or severe pleural adhesions
* Severe adverse reactions
* Severe systemic infection
* With contraindications to the use of electroacupuncture, such as skin damage or infection at the acupoints
* Suffering from nervous system disease or abnormal mental state
* Participate in the other clinical trial 3 month before the enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Dosage of sufentanil used during anesthesia | during the anesthesia
  Dosage of sufentanil used during anesthesia

SECONDARY OUTCOMES:
Evaluation of inotropic scores | 24h postoperatively
  inotropic drugs used postoperatively
Dosage of propofol used during anesthesia | During the anesthesia
  Dosage of propofol used during anesthesia
Time of mechanical ventilation | at 30 days
  length of mechanical ventilation postoperatively
In-hospital stay | at 30 days
  It is the length of hospital stay postoperatively
Incidence of overall complication | at 30 days
  Incidence of overall complication postoperatively
Incidence of overall mortality | at 30 days
  Incidence of overall mortality postoperatively
The length of CCU stay | at 30 days
  Length of CCU stay postoperatively
Heart rate during the anesthesia | during the anesthesia
  Heart rate during the anesthesia
Mean arterial pressure during the anesthesia | during the anesthesia
  Mean arterial pressure during the anesthesia
Bispectral index during the anesthesia | during the anesthesia
  Bispectral index during the anesthesia
Incidence of overall complication | at 1 year
  Incidence of overall complications postoperatively
Incidence of overall mortality | at 1 year
  Incidence of overall mortality postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Li ze Xiong, M.D.,Ph.D., Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China